CLINICAL TRIAL: NCT06613919
Title: Prospective Randomised Trial for 6-Months Versus 9-Months Anti-TB Therapy for Tubercular Posterior Uveitis
Brief Title: Six-months Versus Nine-months ATT for Ocular TB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, HERF, Head, Uveitis Services, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-011-BHR-29
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Tuberculosis (TB); Uveitis; Retinal Vasculitis; Choroiditis
Keywords: Tuberculosis; Uveitis; anti-TB therapy; duration
MeSH Terms: conditions — Tuberculosis; Uveitis; Retinal Vasculitis; Choroiditis

STUDY DESIGN:
Intervention Model Description: Non-inferiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Six months (Experimental): Six months anti-TB therapy
  Interventions: Drug: Anti-Tuberculosis Treatment
- Nine months (Active Comparator): Nine months anti-TB therapy
  Interventions: Drug: Anti-Tuberculosis Treatment

INTERVENTIONS:
Drug: Anti-Tuberculosis Treatment — Standard, weight adjusted anti-TB therapy for six months
  Arms: Six months
Drug: Anti-Tuberculosis Treatment — Standard, weight-adjusted anti-TB therapy for nine months
  Arms: Nine months

SUMMARY:
The goal of this clinical trial is to learn if 6-months anti-TB therapy is not worse than 9-months therapy for the treatment of tubercular posterior uveitis. The main questions it aims to answer are:

Does six-month therapy work as well as the nine-month therapy? Do any of the specific phenotypes of TB posterior uveitis respond better to any specific duration of anti-TB therapy?

Participants:

Took the standard dose of six- or nine-month ATT for TB posterior uveitis Visit the clinic as advised for checkups and tests

DETAILED DESCRIPTION:
1. Tubercular uveitis (TBU) is a major cause of intraocular inflammation in TB-endemic countries. It has several clinical manifestations affecting nearly every tissue in the eye. Histopathological studies of TBU have revealed presence of paucibacillary mycobacterial infection and granulomatous infection in enucleated eyes. Unlike TB in other organ systems, microbiological evidence of TB is rarely found in ocular fluids that are sampled from TBU eyes. Hence, the diagnosis of TBU is based on presence of characteristic clinical signs, ancillary evidence of systemic TB infection and exclusion of non-TB entities. Active pulmonary TB, however, is rarely found in TBU patients.
2. While there are no agreed management guidelines for TBU, several studies, both from TB-endemic and non-endemic countries, have supported the utility of anti-TB therapy (ATT) in the resolution of ocular inflammation, and prevention of recurrence. Delay in initiation of ATT has led to chronic inflammation and prolonged visual impairment in TBU [6]. These studies have typically been retrospective and have included patients with wide range of clinical presentations, based on diagnostic criteria, described above. Majority of these studies have used adjunctive corticosteroids and/or immunosuppressants along with ATT. The duration of ATT in these studies have varied from 6-24 months. A meta-analysis of these studies revealed that 84% (95% CI 79-89) of the patients receiving ATT had no recurrence of inflammation during the follow-up period.

AIM of the study: To compare the efficacy of 6-month with that of 9-month ATT, for the treatment of clinically diagnosed tubercular posterior uveitis (TPU).

Study design: An international, multicenter, prospective, randomized, observer masked-study in three centres spread across India, Myanmar and Thailand.

Patient assesment: This included detailed history of ocular and systemic illnesses, history of TB contact in past, ETDRS best corrected visual acuity (converted from Snellens, if ETDRS unavailable), intraocular pressure by Goldmann applanation tonometry, slit lamp biomicroscopy, and indirect ophthalmoscopy. Fundus photography (seven-field or wide-field, if available) was performed for all patients. Other ocular imaging such as fluorescien angiography, fundus autofluorescence, optical coherence tomography (OCT), OCT-angiography or indocyanine green angiography, were performed as per specific requirements in individual cases. All patients with clinical signs compatible with TPU, were investigated for complete blood counts, erythrocyte sedimentation rate, HIV, VDRL, TST and contrast enhanced computed tomography (CECT) of thorax. If CECT is not available at a centre, then a digital X-ray of the chest was considered in lieu of it. IGRA was performed in conjunction with TST, or in patients with strong suspicion of TPU but negative TST. Additional investigations were performed at the discretion of the investigator to rule out non-TB diagnosis.

Follow-up evaluation were done at 2 weeks, 1 month (+/-1 week), 2 months (+/-2 weeks), 4 months (+/-2 weeks), 6 months (+/-4 weeks), 9 months (+/-4weeks), and then 3 monthly (+/-4 weeks), till one year after completion of ATT. The one-year cut-off limit has been chosen, since most recurrences have been known to occur within one year after the completion of ATT (at least in case of pulmonary TB). Ocular and systemic evaluation, including ocular imaging (as described above), will be performed for each visit.

ELIGIBILITY:
Inclusion Criteria:

* Objective evidence of active intraocular inflammation compatible with TPU e.g. active retinal vasculitis (with FA leakage) or choroidal lesions
* Positive results of tuberculin skin test (TST >=10 mm induration after 48 hours with 5TU) and/or interferon gamma release assay (Quantiferon TB Gold or T-SPOT)
* May have evidence of healed pulmonary or other TB (but not requiring ATT for that disease)
* Age more than 18 years, not pregnant

Exclusion Criteria:

* Ophthalmic findings or ancillary test results consistent with non-TB diagnosis
* Objective findings showing only non-active disease eg. occluded retinal vessels only, with no FA leakage from non-occluded vessels, or atrophic/scarred choroidal lesions
* Optic nerve involvement
* Past history of uveitis
* Previous ATT for ocular or other disease
* Concurrent active pulmonary or other TB disease requiring ATT for that disease.
* HIV infection and other immunocompromised patients
* Treated with systemic or local corticosteroids within 3 months prior to entry
* Received anti-VEGF injections within 3 months prior to entry
* Age <18 years
* Pregnancy
* Liver disease
* Likelihood of poor compliance/ refusal to participate in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Non-recurrence of inflammation | One year after completion of ATT
  Treatment failure after completion of 6- or 9-month ATT.

CONTACTS AND LOCATIONS:
Locations (3):
- University of Medicine Magway, EENT Hospital, Nay Pyi Taw, Burma
- LV Prasad Eye Institute, Bhubaneswar, Odisha, India
- Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
We will need approval from the respective IRBs of each of the three study sites to share the IPD

REFERENCES:
- [Background] Nunn AJ, Phillips PP, Mitchison DA. Timing of relapse in short-course chemotherapy trials for tuberculosis. Int J Tuberc Lung Dis. 2010 Feb;14(2):241-2. PMID 20074418
- [Background] Kee AR, Gonzalez-Lopez JJ, Al-Hity A, Gupta B, Lee CS, Gunasekeran DV, Jayabalan N, Grant R, Kon OM, Gupta V, Westcott M, Pavesio C, Agrawal R. Anti-tubercular therapy for intraocular tuberculosis: A systematic review and meta-analysis. Surv Ophthalmol. 2016 Sep-Oct;61(5):628-53. doi: 10.1016/j.survophthal.2016.03.001. Epub 2016 Mar 10. PMID 26970263